CLINICAL TRIAL: NCT03385551
Title: Observational Study to Evaluate the Acceptability and Efficacy of 10 Micrograms of Estradiol Vaginal Tablets vs Promestriene Vaginal Cream
Brief Title: Study to Evaluate Estradiol Vaginal Tablets vs Promestriene Vaginal Cream
Status: Completed | Type: Observational
Sponsor: Instituto Palacios (Other)
Responsible Party: Sponsor
Other Study IDs: IP-AVV2017
Record Dates: First submitted 2017-11-30; First posted 2017-12-28 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Vulvovaginal Atrophy
Keywords: Vulvovaginal Atrophy
MeSH Terms: interventions — Estradiol; promestriene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ARM 1: Patients who have been prescribed by the physician within the standard clinical practice 10 micrograms of estradiol vaginal tablets. One tablet intravaginally once daily for two weeks. Thereafter one tablet twice per week with at least a 3-days interval between treatments
  Interventions: Drug: Estradiol
- ARM 2: Patients who have been prescribed by the physician within the standard clinical practice promestriene 10mg./g vaginal cream. 1 gr. one application once daily intravaginally for two weeks. Thereafter one application twice per week with at least a 3-days interval between treatments

INTERVENTIONS:
Drug: Estradiol — Estradiol or Promestriene depending on the arm
  Other Names: Promestriene
  Groups: ARM 1

SUMMARY:
This is a study to evaluate the acceptability, efficacy and preferences of 10 of estradiol vaginal tablets vs promestriene vaginal cream

DETAILED DESCRIPTION:
This is an observational, prospective, open-label, parallel-group study to evaluate the acceptability, efficacy, and preferences of postmenopausal women older than 45 between 10 micrograms of estradiol vaginal tablets vs promestriene vaginal cream

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women aged 45 years or older. Women will be considered postmenopausal with more than 12 months since last menstrual period

* Women who have been prescribed vaginal estradiol tablets or vaginal promestriene cream· Women who have read and signed the Informed Consent Form
* Women with an intact uterus
* One or more vaginal symptoms (dryness, soreness, irritation, dyspareunia) rated as moderate to severe. Symptoms are moderate if the patient needs a treatment and feels discomfort. Symptoms are severe if the patient needs a treatment, and feels such a degree of discomfort that this could severely impact the subject's daily activities
* In case of doubt, blood estradiol concentration will be determined, and the subject will only be enrolled if the levels are equal to 30pg./ml. or less.

Exclusion Criteria:

* Women who had a known or suspected history of breast carcinoma

  * Estrogen dependent neoplasia. Women with a known, past or suscpected Estrogen-dependent malignant tumours such as endormetrial or ovarian cancer
  * Positive or suspicious mammogram results
  * Any systemic malignant disease
  * Hormone therapy treatment (sex hormones or vaginal treatments or steroids) in the last three months Women who had abnormal vaginal bleeding or uterine bleeding of unknown cause
  * Vaginal infection requiring treatment
  * Previous or current venous thromboembolism (deep venous thrombosis, pulmonary embolism) Untreated endometrial hyperplasia Known thrombophilic disorders (e.g. protein C, protein S, or antithrombin deficiency) Active or previous arterial thromboembolic disease (e.g. angina, myocardial infarction) Acute liver disease, or history of liver disease as long as liver function tests have failed to return to normal Known Hypersensitivity to the active substances or to any of the excipients Porphyria
  * Any serious disease or chronic condition that could interfere with study compliance
  * History of thrombolytic disorders
  * Use of vaginal contraceptives (DIU, vaginal ring…)
  * Participation in another clinical trial in the last three months.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal Women
Study Population: 120 postmenopausal women aged 45 years or older, with one or more moderate to severe symptoms of vulvovaginal atrophy (dryness, dyspareunia, soreness or irritation)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Vulvovaginal Symptoms | Change from Baseline, at week 4 and at week 12
  Dispareunya, dryness, itching nd burning

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Palacios, MD, Principal Investigator — Instituto Palacios
Locations (2):
- IRCCS "S Matteo Foundation", Pavia, Italy
- Instituto Palacios, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No